CLINICAL TRIAL: NCT03961698
Title: Ph 2, Multi-arm, Multicenter, Open-label Study to Evaluate Efficacy and Safety of IPI-549 Administered in Combo With Front-line Treatment Regimens in Pts With Locally Advanced and/or Metastatic Triple-Negative Breast Cancer or Renal Cell Carcinoma
Brief Title: Evaluation of IPI-549 Combined With Front-line Treatments in Pts. With Triple-Negative Breast Cancer or Renal Cell Carcinoma
Acronym: MARIO-3
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Infinity Pharmaceuticals, Inc. (Industry)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IPI-549-03
Record Dates: First submitted 2019-04-08; First posted 2019-05-23 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Breast Cancer; Renal Cell Carcinoma
Keywords: Phase 2; PI3K; IPI-549; Advanced Solid Tumor; Triple Negative Breast Cancer (TNBC); Renal Cell Carcinoma (RCC); PD-L1; Myeloid-Derived Suppressor Cells (MDSCs); Front-Line Treatment; eganelisib
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Renal Cell; Triple Negative Breast Neoplasms | interventions — IPI-549; atezolizumab; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Bevacizumab

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two or more groups in parallel for the duration of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (TNBC) (Experimental): IPI-549 in combination with front-line treatment. Cohort A will include two sub-cohorts: Cohorts A1 and A2.
  Cohort A1: Approximately 30 patients with locally advanced and/or metastatic TNBC with programmed death-ligand 1 (PDL1) positive disease based on immunohistochemistry (IHC) defined as IC1/2/3.
  Cohort A2: Approximately 30 patients with locally advanced and/or metastatic TNBC with PDL1 negative disease based on IHC defined as IC0.
  Interventions: Drug: IPI-549 (eganelisib); Drug: Atezolizumab; Drug: nab-paclitaxel
- Cohort B (RCC) (Experimental): IPI-549 in combination with front-line treatment. Cohort B will include two sub-cohorts: Cohorts B1 and B2.
  Cohort B1: Approximately 15 patients with locally advanced and/or metastatic RCC, with PDL1 positive disease based on IHC defined as IC1/2/3.
  Cohort B2: Approximately 15 patients with locally advanced and/or metastatic RCC, with PDL1 negative disease based on IHC defined as IC0.
  Interventions: Drug: IPI-549 (eganelisib); Drug: Atezolizumab; Drug: Bevacizumab

INTERVENTIONS:
Drug: IPI-549 (eganelisib) — IPI-549 is an oral, selective inhibitor of phosphoinositide-3-kinase gamma (PI3K-gamma). It is an orally-administered capsule that will be dosed at either 20mg/day, 30mg/day, or 40mg/day to patients in both cohorts A and B depending on the results of the safety run-in phase for each cohort.
Drug: Atezolizumab — Atezolizumab is a fully humanized, engineered monoclonal antibody of IgG1 isotype against the protein programmed cell death-ligand 1 (PD-L1). 840 mg of the drug will be administered intravenously (IV) on days 1 and 15 in combination of each 28-day cycle for patients with TNBC. 1200mg will be administered IV on day 1 of each 21-day cycle to patients with RCC.
  Other Names: Tecentriq
Drug: nab-paclitaxel — Nab-paclitaxel is a nanoparticle albumin-bound formulation of paclitaxel (Taxol), a mitotic inhibitor chemotherapy, with less toxicity than solvent-based (sb) paclitaxel and achieves a 33% higher tumor uptake in preclinical models. Nab-paclitaxel will be administered intravenously (IV) at 100 mg/m2 on days 1, 8 and 15 of each 28-day cycle for patients with TNBC.
  Other Names: Abraxane
  Arms: Cohort A (TNBC)
Drug: Bevacizumab — Bevacizumab is an anti-vascular endothelial growth factor (anti-VEGF) recombinant monoclonal antibody that is approved by the FDA for the treatment of multiple solid tumors in combination with chemotherapy. It will be administered at 15 mg/kg IV on day 1 of each 21-day cycle to patients with RCC.
  Other Names: Avastin
  Arms: Cohort B (RCC)

SUMMARY:
MARIO-3 is a Phase 2 multi-arm combination cohort study designed to evaluate IPI-549, Infinity Pharmaceutical's first-in-class, oral immuno-oncology product candidate targeting immune-suppressive tumor-associated myeloid cells through selective inhibition of phosphoinositide-3-kinase (PI3K)-gamma, in combinations with Tecentriq and Abraxane (nab-paclitaxel) in front-line triple negative breast cancer (TNBC) and in combination with Tecentriq and Avastin (bevacizumab) in front-line renal cell cancer (RCC).

DETAILED DESCRIPTION:
MARIO-3 (Macrophage Reprogramming in Immuno-Oncology) is a prospective Phase 2 multi-arm, multicenter, open-label, combination cohort study designed to evaluate IPI-549, Infinity Pharmaceutical's first-in-class, oral immuno-oncology product candidate targeting immune-suppressive tumor-associated myeloid cells through selective inhibition of phosphoinositide-3-kinase (PI3K)-gamma. IPI-549 will be administered in combinations with Tecentriq and Abraxane (nab-paclitaxel) in front-line triple negative breast cancer (TNBC) and in combination with Tecentriq and Avastin (bevacizumab) in front-line renal cell cancer (RCC).

This study will enroll approximately 90 treatment-naïve patients across the following disease cohorts. Cohort A will be composed of patients with locally advanced and/or metastatic triple-negative breast cancer (TNBC). Cohort B will be composed of patients with locally advanced and/or metastatic renal cell carcinoma (RCC).

The primary objective of MARIO-3 is to evaluate the complete response (CR) rate per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 following combination treatment with IPI-549 and front-line treatment in patients with TNBC and RCC. Its secondary objectives include evaluation of the safety, objective response rate (ORR), time to CR (TTCR), time to response (TTR), duration of CR (DOCR), duration of response (DOR), and progression-free survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age.
2. Have signed and dated an independent review board (IRB)/independent ethics committee (IEC) approved informed consent form (ICF) in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol-related procedures that are not part of normal patient care.
3. Willing and able to comply with scheduled visits, treatment schedule, laboratory tests, fresh tumor biopsies, and all other protocol requirements.
4. At least 1 measurable disease lesion by computed tomography (CT) or magnetic resonance imaging (MRI) as defined by RECIST v1.1 performed within 1 week prior to first dose.
5. Willing to undergo one pre-treatment core biopsy (unless archival tumor tissue is available within 3 months of first dose) and one on-treatment tumor biopsy, unless not safe or medically feasible. If the patient is unwilling to undergo biopsy, they may be eligible with approval of the medical monitor.
6. Evaluable tumor tissue (archived [without time constraints] or new biopsy) must be provided for biomarker analysis, which will include PD-L1 expression level using immunohistochemistry (IHC) to measure specific PD-L1 signals in tumor-infiltrating immune cells (ICs). Results are not required prior to start of study treatment.
7. Eastern Cooperative Oncology Group (ECOG) performance status ≤1.
8. Life expectancy ≥12 weeks.
9. Baseline laboratory values must meet the following criteria within 14 days of the first dose:

   1. Adequate hematologic function, defined as white blood cell (WBC) count ≥2.0 × 109/L, absolute neutrophil count ≥1.5 × 109/L (without granulocyte colony-stimulating factor [GCSF] support within 2 weeks prior to Cycle 1, Day 1), lymphocyte count ≥0.5 × 109/L, hemoglobin ≥9.0 g/dL (patients may be transfused or receive erythropoietic treatment to meet this criterion), and platelet count ≥100 × 109/L (without transfusion within 2 weeks prior to Cycle 1, Day 1).
   2. Calculated creatinine clearance ≥30 mL/min.
   3. Aspartate aminotransferase (AST), alanine aminotransferase (ALT) and alkaline phosphatase (ALP) <2.5 × upper limit of normal (ULN). ALT and AST ≤5 × ULN if documented liver metastasis. ALP ≤5 × ULN if documented bone or liver metastasis.
   4. Total bilirubin ≤1.25 × ULN (unless elevated due to Gilbert's syndrome who can have total bilirubin <3.0 mg/dL).
   5. International normalized ratio (INR) and activated partial thromboplastin time (aPTT) ≤1.5 × ULN. This applies to patients who are not receiving therapeutic anticoagulation; patients receiving therapeutic anticoagulation should be on a stable dose.
   6. Serum albumin >2.5 g/dL
10. Women of childbearing potential (WOCBP) must have a negative serum or urine β human chorionic gonadotropin (βhCG) pregnancy test within 1 week before administration of study drug WOCBP is defined as any female who has ≥12 months of non-therapy induced amenorrhea or is surgically sterile.
11. Women must not be breastfeeding.
12. Willingness of male and female patients who are not surgically sterile or postmenopausal to use medically acceptable methods of birth control for the duration of study treatment, including 30 days after the last dose of IPI-549 and of nab-paclitaxel, or 6 months after the last dose of atezolizumab or bevacizumab, whichever is later. Male patients must refrain from donating sperm for these same periods. Male patients with a pregnant female partner must agree to remain abstinent or use a condom during the treatment period and for the duration of the pregnancy.

Patients in Cohort A must meet the following additional criteria for inclusion:

1. Women with metastatic or locally advanced (not amenable to resection with curative intent), histologically documented TNBC, i.e., absence of human epidermal growth factor receptor 2 (HER2), estrogen receptor (ER) and progesterone receptor (PR) expression:

   1. HER2 negativity defined as either of the following by local laboratory assessment
   2. ER and PR negativity defined as <1% of cells expressing hormonal receptors via IHC analysis
2. No prior chemotherapy or targeted systemic therapy for inoperable locally advanced or metastatic TNBC. Radiation therapy for metastatic disease is permitted. There is no required minimum washout period for radiation therapy. Patients should be recovered from the effects of radiation. Prior chemotherapy (including taxanes) in the neoadjuvant or adjuvant setting is allowable if treatment was completed ≥12 months prior to randomization.

Patients in Cohort B must meet the following additional criteria for inclusion:

1. Men or women with histologically documented unresectable advanced or metastatic RCC with clear-cell histology.
2. No prior treatment with active or experimental systemic agents, including treatment in the neoadjuvant or adjuvant setting. Prior radiotherapy is permitted but must not have been administered within 14 days of Cycle 1, Day 1.

Exclusion Criteria:

1. WOCBP who are pregnant or breastfeeding.
2. Women with a positive pregnancy test at enrollment or prior to administration of study medication.
3. Any serious or uncontrolled medical disorder that, in the opinion of the Investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the patient to receive protocol therapy, or interfere with the interpretation of study results, including significant liver disease (such as cirrhosis, uncontrolled major seizure disorder, or superior vena cava syndrome).
4. Any history of, or currently active, brain or leptomeningeal metastases.
5. Significant cardiovascular disease, such as New York Heart Association (NYHA) cardiac disease (Class II or greater), myocardial infarction within 3 months prior to randomization, unstable arrhythmias, or unstable angina. Patients with a known left ventricular ejection fraction (LVEF) <40% will be excluded. Patients with known coronary artery disease, congestive heart failure not meeting the above criteria, or LVEF <50% must be on a stable medical regimen that is optimized in the opinion of the treating physician, in consultation with a cardiologist if appropriate.
6. Baseline QT interval corrected with Fridericia's method (QTcF) >480 ms.
7. Major surgical procedure within 4 weeks prior to enrollment or anticipation of the need for a major surgical procedure during the course of the study other than for diagnosis. Placement of central venous access catheter(s) (e.g., port or similar) is not considered a major surgical procedure and is therefore permitted.
8. Active tuberculosis.
9. Ongoing systemic bacterial, fungal, or viral infections at Screening.
10. Positive test for human immunodeficiency virus (HIV).
11. Active hepatitis B (defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) or hepatitis C. Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen [anti-HBc] antibody test) are eligible. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
12. Dependence on continuous supplemental oxygen use.
13. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently). Patients with indwelling catheters (e.g., PleurX®) are allowed.
14. Uncontrolled hypercalcemia (>1.5 mmol/L ionized calcium or calcium >12 mg/dL or corrected serum calcium >ULN) or symptomatic hypercalcemia requiring continued use of bisphosphonate therapy. Patients who are receiving denosumab must discontinue denosumab use and replace it with a bisphosphonate instead while on study. There is no required minimum washout period for denosumab. Patients who are receiving bisphosphonate therapy specifically to prevent skeletal events and who do not have a history of clinically significant hypercalcemia are eligible.
15. Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells, or any of the study drug components.
16. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins.
17. History of stroke, transient ischemic attack, or ventricular arrhythmia requiring medication or mechanical control within the last 6 months prior to Screening.
18. Other prior malignancy active within the previous 5 years except for local or organ confined early stage cancer that has been definitively treated with curative intent, does not require ongoing treatment, has no evidence of residual active disease, and has a negligible risk of recurrence and is therefore unlikely to interfere with the primary and secondary endpoints of the study, including response rate and safety.
19. History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis.
20. History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest CT scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
21. Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease.
22. Prior allogeneic stem cell or solid organ transplantation.
23. Administration of a live or attenuated vaccine within 4 weeks of first dose of study drug or anticipation that such a live or attenuated vaccine will be required during the study or within 5 months following the last dose of atezolizumab.
24. Prior therapy with experimental anti-tumor vaccines; any T cell co-stimulation or checkpoint pathways, such as anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody, including ipilimumab, or other medicines specifically targeting the T cell; or IPI-549.
25. Treatment with systemic immunostimulatory agents (including but not limited to interferons or IL-2) within 4 weeks or 5 half-lives of the drug (whichever is shorter) prior to enrollment.
26. Treatment with systemic corticosteroids or other systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [TNF] agents) within 2 weeks prior to randomization, or anticipated requirement for systemic immunosuppressive medications during the trial.
27. Treatment with botanical preparations (e.g., herbal supplements or traditional Chinese medicines) intended for general health support or to treat the disease under study within 2 weeks prior to randomization.
28. Administration of any of the following within 1 week prior to the administration of study drug:

    1. Strong inhibitors or inducers of cytochrome P450 (CYP) 3A4, including grapefruit, grapefruit juice and herbal supplements.
    2. Warfarin, phenytoin, or other substrates of CYP2C8 or CYP2C9 with a narrow therapeutic range.
    3. P-glycoprotein (P-gp) inhibitors.
29. Prior surgery or gastrointestinal dysfunction that may affect drug absorption (e.g., gastric bypass surgery, gastrectomy).

Patients in Cohort A are to be excluded from the study if they meet any of the following criteria:

1. Spinal cord compression not definitively treated with surgery and/or radiation, or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for >2 weeks prior to first dose of study treatment.
2. Uncontrolled tumor-related pain.
3. Known hypersensitivity to nab-paclitaxel or to any of the excipients.

Patients in Cohort B are to be excluded from the study if they meet any of the following criteria:

1. Inadequately controlled hypertension (systolic blood pressure >150 mmHg and/or diastolic blood pressure >100 mmHg or prior history of hypertensive crisis or hypertensive encephalopathy.
2. Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Cycle 1, Day 1.
3. Evidence of bleeding diathesis or clinically significant coagulopathy (in the absence of therapeutic anticoagulation).
4. Current or recent (within 10 calendar days prior to Cycle 1, Day 1) use of dipyridamole, clopidogrel, or cilostazol.
5. History of abdominal or tracheoesophageal fistula or gastrointestinal perforation within 5 months prior to Cycle 1, Day 1.
6. Clinical signs or symptoms of gastrointestinal obstruction or requirement for routine parenteral hydration, parenteral nutrition, or tube feeding.
7. Evidence of abdominal free air not explained by paracentesis or recent surgical procedure.
8. Serious, non-healing or dehiscing wound, active ulcer, or untreated bone fracture.
9. Proteinuria, as demonstrated by urine dipstick or >1.0 g of protein in a 24-hour urine collection. All patients with ≥2+ protein on dipstick urinalysis at baseline must undergo a 24-hour urine collection for protein.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Complete Response (CR) rate (change in target lesion size). | CR rate assessments will be conducted through month 12 for Cohort A (TNBC) and through month 18 for Cohort B (RCC) until unacceptable toxicity, confirmed progression of disease, withdrawal of consent, or other treatment discontinuation criteria are met.
  Complete Response (CR) rate is defined per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 as disappearance of all target and non-target lesions.

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | TEAE assessments will be conducted from screening through month 12 for Cohort A (TNBC) and from screening through month 18 for Cohort B (RCC). Additional assessments will be conducted 30 days and 90 days from last dose.
  Treatment emergent adverse events (TEAE) are undesirable events not present prior to medical treatment, or an already present event that worsens either in intensity or frequency following the treatment.
Incidence of serious adverse events (SAEs), including deaths | SAE assessments will be conducted from screening through month 12 for Cohort A (TNBC) and from screening through month 18 for Cohort B (RCC). Additional assessments will be conducted 30 days and 90 days from last dose.
  Serious adverse events include death, life-threatening events, initial or prolonged hospitalization, disability or permanent damage, or require an intervention to prevent impairment.
Incidence of adverse events (AEs) leading to treatment discontinuation | AE assessments will be conducted from screening through month 12 for Cohort A (TNBC) and from screening through month 18 for Cohort B (RCC). Additional assessments will be conducted 30 days and 90 days from last dose.
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An adverse event (AE) can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Changes from baseline in electrocardiograms (ECGs) | ECG assessments will be performed from screening through month 12 for Cohort A (TNBC) and from screening through month 18 for Cohort B (RCC).
  ECGs assess heart problems by measuring the electrical activity generated by the heart as it contracts. The components that will be assessed during the ECG are P wave, QRS complex, ST segment, and T wave.
Objective response rate (ORR) | ORR will be assessed from screening through month 12 for Cohort A (TNBC) and from screening through month 18 for Cohort B (RCC).
  ORR is defined as best response of CR or partial response (PR), as determined by RECIST v1.1.
Time to Complete Remission (TTCR) | TTCR will be assessed from screening through month 12 for Cohort A (TNBC) and from screening through month 18 for Cohort B (RCC).
  TTCR is defined as the time from the first dose of study treatment to CR.
Time to response (TTR) | TTR will be assessed from screening through month 12 for Cohort A (TNBC) and from screening through month 18 for Cohort B (RCC).
  TTR is defined as the time from the first dose of study treatment to first objective response (CR or PR) in patients with CR or PR.
Duration of Complete Remission (DOCR) | DOCR will be assessed from screening through month 12 for Cohort A (TNBC) and from screening through month 18 for Cohort B (RCC).
  DOCR is defined as the time from the first CR to documented disease progression in patients with CR.
Duration of response (DOR) | DOR will be assessed from screening through month 12 for Cohort A (TNBC) and from screening through month 18 for Cohort B (RCC).
  DOR is defined as the time from the first objective response (CR or PR) to documented disease progression in patients with CR or PR.
Progression-free survival (PFS) | PFS will be assessed from screening through month 12 for Cohort A (TNBC) and from screening through month 18 for Cohort B (RCC).
  PFS is defined as the time from the first dose of study treatment to documented disease progression or death due to any cause.
Population Pharmacokinetics (PK) of IPI-549 | PK assessments will be performed on day 1 of each 28-day cycle through cycle 2 for cohort A (TNBC) at and on day 1 of each 21-day cycle through cycle 2 for cohort B (RCC).
  Population PK estimates (variability in drug concentrations within the study population measured in ng/mL) includes inter- and intra-subject variability and covariate effects.
Pharmacokinetics (PK) of Atezolizumab | PK assessments will be performed on day 1 of cycle 1, on day 1 of cycles 2 through 4, C8D1, C16D1 for both cohorts. Cohort A (TNBC) has a 28-day cycle and cohort B (RCC) has a 21-day cycle.
  Concentration of Atezolizumab in the blood at predose measured in ug/mL.
Changes from baseline in pulse rate | Pulse rate will be assessed from screening through month 12 for Cohort A (TNBC) and from screening through month 18 for Cohort B (RCC).
  Pulse rate as measured in beats per minute (bpm).
Changes from baseline in temperature | Temperature will be assessed from screening through month 12 for Cohort A (TNBC) and from screening through month 18 for Cohort B (RCC).
  Temperature as measured in celsius.
Changes from baseline in respiration rate | Respiration rate will be assessed from screening through month 12 for Cohort A (TNBC) and from screening through month 18 for Cohort B (RCC).
  Respiration rate as measured in breaths per minute.
Changes from baseline in blood pressure | Blood pressure will be assessed from screening through month 12 for Cohort A (TNBC) and from screening through month 18 for Cohort B (RCC).
  Systolic and diastolic blood pressure as measured in mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Feng Chi, PhD, RN, Study Director — Medical Lead
Locations (24):
- United States (24):
  - Ironwood Cancer and Research Center, Chandler, Arizona
  - Arizona Oncology Associates, Tucson, Arizona
  - Arizona Clinical Research Center, Tucson, Arizona
  - St. Joseph Heritage Healthcare, Fullerton, California
  - Cancer & Blood Specialty Clinic, Los Alamitos, California
  - Sharp Memorial Hospital, San Diego, California
  - Samsum Clinic, Santa Barbara, California
  - UCLA, Santa Monica, California
  - Olive View - UCLA Medical Center, Sylmar, California
  - Valley Breast Cancer Care and Women's Health Center, Van Nuys, California
  - University of Colorado, Aurora, Colorado
  - Orlando Health, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - University Cancer & Blood Center, Athens, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Cancer Center of Kansas, Wichita, Kansas
  - Norton Cancer Institute, Louisville, Kentucky
  - University of Maryland, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Tennessee Oncology, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - UT Health East Texas HOPE Cancer Center, Tyler, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: IPI-549 — http://www.infi.com/home/our-development-program/ipi-549/